CLINICAL TRIAL: NCT06689735
Title: Investigation of the Effectiveness of Schroth Exercises and Pilates Exercises in Patients With Scoliosis: A Randomized Trial
Brief Title: Investigation of the Effectiveness of Schroth Exercises and Pilates Exercises in Patients With Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar15
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Scoliosis
MeSH Terms: conditions — Scoliosis | interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Schroth (Experimental): 3D corrective scoliosis exercises
  Interventions: Other: schroth exercises
- Pilates (Experimental): Pilates exercises
  Interventions: Other: pilates exercises

INTERVENTIONS:
Other: schroth exercises — Exercises will be given in lying, sitting and standing positions. In each exercise, elongation of the spine will be ensured and the person will be positioned according to the type of scoliosis. Exercises will be given progressively in supine, prone, side sitting, sitting and standing positions. In each exercise, elongation of the spine will be ensured and the person will be positioned according to the upper and lower extremities. Progress in the exercises will be made positionally by increasing the number of repetitions and the number of rotational breathing during the exercise.
  Arms: Schroth
Other: pilates exercises — The average application time of the exercises is 30-40 minutes (with the first 10 minutes of warming up and the last 5 minutes of stretching). The first four exercises were used for the warm-up period and the last four exercises were used for the stretching period. The exercises will be done as 1 set of 8 repetitions. The Hundred exercise will be increased to 10 sets of 10 reps every two weeks to 10 reps, 12 reps, and 14 reps, respectively.
  Arms: Pilates

SUMMARY:
The aim of this study is to examine the effectiveness of Schroth exercises and Pilates exercises in patients with scoliosis.

DETAILED DESCRIPTION:
The study was planned as a randomized controlled trial. The randomization process will be done as block randomization using the random interval command in Microsoft Excel. The participants to be included in the study will be selected from the clients receiving consultancy services at the Mehmet Gümüş (MG) Clinic Physiotherapy and Wellness Center. 50 individuals diagnosed with scoliosis who applied with a postural disorder complaint will be included in the study. The individuals will be randomly divided into 2 equal groups. The rehabilitation program of the 25 individuals in the first group will be planned as 3-dimensional corrective scoliosis exercises. The program of the 25 individuals in the second group will be applied as pilates scoliosis exercises. After the initial evaluations explained to the individuals included in the study are made, an exercise program of a total of 36 sessions, each lasting approximately 50 minutes, will be applied by experienced physiotherapists who have received 3-dimensional exercise method training and pilates training specific to scoliosis, 3 days a week for 12 weeks.

ELIGIBILITY:
INCLUSION CRITERIA:

* Being between 18-45 years of age
* Having a primary curve between 10-40 degrees according to the Cobb method
* Having typical S or C scoliosis
* Being willing to participate in the study
* Having the cognitive capacity to cooperate with the guidance of a physiotherapist
* EXCLUSION CRITERIA:
* Having a BMI over 30 kg/m²
* Having any neurological, orthopedic, cardiopulmonary disorders other than the diagnosis of scoliosis
* Having any injuries related to the musculoskeletal system in the last 6 months
* Being unable to fulfill exercise requirements for any reason

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
The Pittsburgh Sleep Quality Index (PSQI) | 14 weeks
  Pittsburgh Sleep Quality Index; It evaluates sleep duration, sleep disturbance, sleep efficiency, subjective sleep quality, sleep medication use, daytime dysfunction, and sleep delay and consists of a total of 24 questions. 19 of them are self-report scales and 5 of them consist of questions to be answered by a friend or spouse. There are 7 components with 18 questions scored in the scale, and each component is evaluated between 0 and 3 points. The total score ranges from 0 to 21, and 5 or more is an indicator of "poor sleep quality".
Scoliosis Research Society-22 | 14 weeks
  Scoliosis Research Society-22 is a functional survey for the patient to fill out on their scoliosis. This survey has been validated in the literature. It is a 22 question survey on the functional status and pain that a patient experiences. Created by the scoliosis research society. There is a scoring rubric that goes with the survey. This survey has 5 domains that are covered with the minimum score of 22 and the maximum score of 110. The higher the score the better the patient is doing in the domains of: Activities of Daily Living, Mental Health, Pain, Patient Satisfaction, Positive Affect, Quality of Life, Social Relationships, and Stress/Coping.
Scoliometer Degree | At time of enrollment
  The degree of rotation measured clinically with a scoliometer
Walter Reed Visual Assessment Scale | 14 weeks
  Walter Reed Visual Assessment Scale (WRGDS) is an evaluation scale created from visual figures. It was developed by Pineda et al. in 2006, for use in individuals with scoliosis, to measure how a person thinks about the deformity in their own body and how severe it is perceived.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Ali Gümüş, Study Chair — Uskudar University; Berna Karamancıoğlu, M.Sc., Study Chair — Uskudar University; Beyzanur Dikmen Hoşbaş, M.Sc., Study Chair — Uskudar University
Locations (1):
- MG Clinic, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karavidas N, Iakovidis P, Chatziprodromidou I, Lytras D, Kasimis K, Kyrkousis A, Apostolou T. Physiotherapeutic Scoliosis-Specific Exercises (PSSE-Schroth) can reduce the risk for progression during early growth in curves below 25 degrees : prospective control study. Eur J Phys Rehabil Med. 2024 Apr;60(2):331-339. doi: 10.23736/S1973-9087.24.08177-2. Epub 2024 Mar 19. PMID 38502554
- [Background] Manzak Dursun AS, Ozyilmaz S, Ucgun H, Elmadag NM. The effect of Pilates-based exercise applied with hybrid telerehabilitation method in children with adolescent idiopathic scoliosis: A randomized clinical trial. Eur J Pediatr. 2024 Feb;183(2):759-767. doi: 10.1007/s00431-023-05340-2. Epub 2023 Nov 23. PMID 37993666
- [Background] Zhang P, Shen X, Zhang L, Wang S, Wu Q. Effect of sling exercise combined with Schroth therapy on adolescents with mild idiopathic scoliosis: A twelve-week randomized controlled trial. J Back Musculoskelet Rehabil. 2024;37(2):379-388. doi: 10.3233/BMR-230102. PMID 38043003